CLINICAL TRIAL: NCT04923243
Title: The Neuro-epigenetics Biomarkers of Postoperative Delirium in Elderly Patients Undergoing Hip/Knee Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HBRC202004072021014
Record Dates: First submitted 2021-04-20; First posted 2021-06-11 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium group: Group of patients with postoperative delirium
  Interventions: Procedure: hip/knee replacement
- Non delirium group: Group of patients without postoperative delirium
  Interventions: Procedure: hip/knee replacement

INTERVENTIONS:
Procedure: hip/knee replacement — hip/knee replacement

SUMMARY:
Introduction: Postoperative delirium (POD), an acute, transient, fluctuating disturbance in attention, cognition, and level of consciousness, is a common (15-53%) postoperative complication, and it is associated with longer hospital stays, worse functional outcomes, higher healthcare costs, and increased mortality. However, at the current time, effective prevention and treatment are not only hampered by lack of knowledge about the neuropathogenesis of POD but also by a lack of biomarkers that could predict individual risk and assess diagnosis and severity of POD.

Recent studies have focused on inflammatory markers (IL-1, IL-6, IL-8, IL-10, CRP), Alzheimer's disease-related factors (Tau, Aβ40/42), and nerve injury factors (S100β, NSE), but failed to establishing causality between these markers and POD. Furthermore, these results were contradictory. Previous study of the investigators found that the dysregulation of preoperative microRNA (miR)-146a and miR-181c in cerebrospinal fluid (CSF) and serum was associated with the development and severity of POD. Therefore, the investigators hypothesized these neurimmiRs and other neuro-epigenetics biomarkers might participate in the neuropathogenesis of POD.

Purpose: Aims to search for neuro-epigenetics biomarkers to predict and diagnose POD.

DETAILED DESCRIPTION:
Method:

1. Study design: This study is a prospective investigation that searches for neuro-epigenetics biomarkers to predict and diagnose POD.
2. Inclusion criteria / Exclusion Criteria

Inclusion criteria: Eligible patients were at least 65 years old and were scheduled to have hip/knee replacement.

Exclusion Criteria:

1. a past medical history of neurological or clinically evident neurovascular disease (e.g., Alzheimer's disease, other forms of dementia, stroke);
2. Patients diagnosed with malignant or benign tumors;
3. Mini-Mental State Examination (MMSE) scores of 26 or less;
4. American Society of Anesthesiologists (ASA) score [a global score that assesses the physical status of patients before surgery, ranging from 1 (normal health) to 5 (moribund)] greater than 3;
5. a history of alcohol abuse and drug dependence;
6. inability to read or severe visual or auditory deficits;
7. unwillingness to comply with the protocol or procedures.

ELIGIBILITY:
Inclusion Criteria: Eligible patients were at least 65 years old and were scheduled to have hip/knee replacement.

Exclusion Criteria:

1. a past medical history of neurological or clinically evident neurovascular disease (e.g., Alzheimer's disease, other forms of dementia, stroke);
2. patients diagnosed with malignant or benign tumors;
3. Mini-Mental State Examination (MMSE) scores of 26 or less;
4. American Society of Anesthesiologists (ASA) score greater than 3;
5. a history of alcohol abuse and drug dependence;
6. inability to read or severe visual or auditory deficits;
7. unwillingness to comply with the protocol or procedures.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were at least 65 years old and were scheduled to have hip/knee replacement.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
cell-free DNA, cell-free RNA and exosomal RNA level in blood and urine | just before surgery
  Cell-free DNA, cell-free RNA and exosomal RNA level in blood and urine of the participants were measured by DNA sequencing or RNA sequencing before surgery.
genome-specific difference between POD and non-POD patients | just before surgery
  Compare the exon sequence in blood samples of the participants, as assessed by whole exome sequencing.
candidate cell-free DNA, cell-free RNA and exosomal RNA level in blood and urine | post operative day 1
  Candidate cell-free DNA, cell-free RNA and exosomal RNA identified in the first outcome were quantified by PCR or RT-PCR on post operative day 1.
candidate cell-free DNA, cell-free RNA and exosomal RNA level in blood and urine | post operative day 3
  Candidate cell-free DNA, cell-free RNA and exosomal RNA were quantified by PCR or RT-PCR on post operative day 3.
candidate cell-free DNA, cell-free RNA and exosomal RNA level in blood and urine | post operative day 7 or the day after delirium disappeared
  Candidate cell-free DNA, cell-free RNA and exosomal RNA were quantified by PCR or RT-PCR on post operative day 7 or the day after delirium disappeared.

SECONDARY OUTCOMES:
Delirium assessment - 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) | before surgery (from 1 week before to the day before)
  positive or negative
Delirium assessment - 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) | post operative day 1
  positive or negative
Delirium severity assessment - Delirium Severity based on 3D-CAM (3D-CAM-S) | post operative day 1
  ranging from 0 to 7 points
Delirium subtype assessment - Richmond Agitation-Sedation Scale (RASS) | post operative day 1
  ranging from -5 to +4 points
Delirium assessment - 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) | post operative day 3
  positive or negative
Delirium severity assessment - Delirium Severity based on 3D-CAM (3D-CAM-S) | post operative day 3
  ranging from 0 to 7 points
Delirium subtype assessment - Richmond Agitation-Sedation Scale (RASS) | post operative day 3
  ranging from -5 to +4 points
Delirium assessment - 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) | post operative day 7 or the day after delirium disappeared
  positive or negative
Delirium severity assessment - Delirium Severity based on 3D-CAM (3D-CAM-S) | post operative day 7 or the day after delirium disappeared
  ranging from 0 to 7 points
Delirium subtype assessment - Richmond Agitation-Sedation Scale (RASS) | post operative day 7 or the day after delirium disappeared
  ranging from -5 to +4 points

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No